CLINICAL TRIAL: NCT06195605
Title: Investigating Age Dependence of Fibroblast and Extracellular Matrix Responses to Cross-linked Hyaluronic Acid Filler in Human Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Gary Fisher, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00230920
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Photoaging
Keywords: Extracellular matrix; Hyaluronic acid; dermal filler
MeSH Terms: interventions — Pharmaceutical Vehicles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Photodamaged skin (Experimental)
  Interventions: Device: Restylane-L; Device: Vehicle

INTERVENTIONS:
Device: Restylane-L — Using a small gauge metal hub needle, two injections of CL-HA dermal filler (Restylane-L) will be performed, each into a small area (approximately 2 x 2 cm) of the mid-dermis of a forearm of a subject. Each injection will be 0.5 cc in volume, and will be approximately 2 cm apart from each other
Device: Vehicle — Two injections of vehicle will be performed in the same manner as Restylane-L and in the same forearm, totaling 4 injections. A plastic template will be used to track the location of the injections, relative to landmarks on the skin.

SUMMARY:
The purpose of the study is to investigate the impact of the injection of dermal filler on the quality of the skin dermal extracellular matrix in persons between the ages of 30-50 years. The quality of the dermal extracellular matrix will be assessed following injection of dermal filler compared to injection of saline vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must understand and sign the informed consent prior to participation
* Subjects must be in generally good health
* Subjects must be able and willing to comply with the requirements of the protocol

Exclusion Criteria:

* Pregnant, plan to become pregnant during the study, or are nursing a child. Participants will be asked to self-report pregnancy
* Individuals with bleeding disorders
* Tend to heal poorly or form very thick scars called keloids
* Have a lidocaine sensitivity, including those with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.
* Individuals with active inflammation or infection of the skin, including active herpes infection.
* Have a significant medical history or concurrent condition which the investigator(s) feel is not safe for study participation, including history of frequent herpes infections, and subjects planning to be exposed to excessive sun, Ultraviolet lamps and extreme cold weather during the first week after injection.
* History of allergies to gram positive bacterial proteins
* Individuals with who have undergone therapy with thrombolytics, anticoagulants, or inhibitors of platelet aggregation in the preceding 3 weeks.
* Have an active inflammation or infection of the skin near the site of injection
* Are taking any medications that suppress your immune system
* Have severe allergies to medications or other things that we believe might make participation unsafe for you
* Have a history of connective tissue diseases, such as:

  * rheumatoid arthritis
  * scleroderma
  * polymyositis/dermatomyositis
  * systemic lupus erythematosus (SLE)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Extracellular Matrix (ECM) deposition as measured using histological stain(s) of skin | Approximately 4 weeks
  Reported as a semi-quantitative grade. The grading scale is 1-4. The higher the number to increased ECM deposition.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fisher, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No